CLINICAL TRIAL: NCT02751866
Title: Early Intervention in Cognitive Aging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Robert Krikorian, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015-1256
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Overweight, Obesity and Other Hyperalimentation (E65-E68)
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Intervention with carbohydrate restriction designed to produce adaptation to ketone metabolism OR intervention with berry fruit powder supplementation.
Who Masked: Participant, Investigator
Masking Description: There is no blind in the dietary intervention given that participants are aware of the nature of the foods they consume. However, each dietary approach is described as healthy. In the berry supplementation studies, there is double blinding using berry fruit and placebo powders that are packaged with a code.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active supplement, low carbohydrate (Active Comparator): Whole fruit berry powder, low carbohydrate diet
  Interventions: Dietary Supplement: Berry fruit powder OR nutritional ketosis
- Placebo, Control (Placebo Comparator): placebo powder, higher carbohydrate diet
  Interventions: Dietary Supplement: Placebo powder OR higher carbohydrate

INTERVENTIONS:
Dietary Supplement: Berry fruit powder OR nutritional ketosis — Daily supplementation with berry fruit powder OR carbohydrate restriction to achieve nutritional ketosis
  Arms: Active supplement, low carbohydrate
Dietary Supplement: Placebo powder OR higher carbohydrate — Daily supplementation with placebo powder OR higher carbohydrate intake
  Arms: Placebo, Control

SUMMARY:
Nutritional intervention in overweight middle aged individuals with subjective memory complaints.

DETAILED DESCRIPTION:
Late-onset AD develops over many years during a preclinical period in which neuropathological changes accumulate before dementia is evident. Deposition of amyloid-beta (Aβ) in the brain is the earliest recognized biomarker of AD pathology, and, demographically, Aβ accumulation begins to accelerate at age 50, a period when the incidence of metabolic disturbance increases as well. Hyperinsulinemia associated with insulin receptor resistance has been associated with AD pathololgy, and metabolic disturbance in mid-life increases risk for subsequent dementia. There are indications that subjective memory complaints can be an early indicator of developing neuropathology and may be the first manifestation of future dementia. This research involves intervention studies in different samples of individuals from this population to investigate the extent to which berry fruit supplementation and ketone metabolism might improve cognitive performance in association with enhancement of metabolic function and related factors. The ultimate goal of this research is to develop interventional approaches that might be applied with at-risk individuals in the preclinical period of dementia to forestall or prevent progression of neurocognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* overweight; subjective memory complaints

Exclusion Criteria:

* diabetes; liver or kidney disease; age-related memory disorder; neurologic or psychiatric condition; substance abuse

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | Eight or 12 weeks after enrollment
  HOMA-IR will be derived from fasting glucose and insulin
Cognitive function | Eight or 12 weeks after enrollment
  Performances on examiner-adminstered instruments assessing memory function

SECONDARY OUTCOMES:
Long term glucose concentration | Eight or 12 weeks after enrollment
  Glycated hemoglobin value

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krikorian, PhD, Principal Investigator — University of Cincinnati Academic Health Center
Locations (1):
- Dept of Psychiatry & Behavioral Neuroscience, UC Academic Health Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No